CLINICAL TRIAL: NCT05385315
Title: Evaluation De La Performance Clinique D'un Nouveau Biomarqueur Sanguin Des Phases Précoces De La Maladie De Parkinson
Brief Title: Towards the Validation of a New Blood Biomarker for the Early Diagnosis of Parkinson's Disease
Acronym: BIOPARK
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Grenoble Institut des Neurosciences (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.0421; 2022-A00337-36 (Other: ID RCB)
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Parkinson's Disease, de novo: patients with de novo PD, without dopaminergic treatment
- Parkinson's Disease, advanced stage: PD patients with diagnosis >5years, with dopaminergic treatment and motor fluctuations.
- Multiple system atrophy: patients with multiple system atrophy

SUMMARY:
The investigators have recently discovered a metabolic biomarker which predicts Parkinson's disease (PD) at the early stages in patients and in animal models. The aim of BIOPARK is to investigate how the biomarker evolves in advanced PD stage, when diagnosis confirmation is higher, an in de novo PD patients who come from a different geographical area than those of the publication (since it is known that the metabolome is largely influenced by lifestyle). They will also evaluate if the biomarker is able to distinguish patients with a parkinsonian syndrome often confused with parkinson's disease, i.e. Multiple System Atrophy (MSA).

DETAILED DESCRIPTION:
Parkinson's disease (PD) affects more than 7 million people worldwide and represents a growing health and socio-economic burden. It is an incurable neurodegenerative disease, and the search for biomarkers that allow reliable early diagnosis and provide new therapeutic targets is essential to find cures for PD.

In a recently published preclinical and clinical study, the investigators have identified in 2 rat models of PD and a primate model and in 2 human cohorts from biobanks significant deregulations of 6 serum metabolites: acetoacetate, betaine, beta-hydroxybutyrate, creatine, pyruvate and valine. From these 6 metabolites, they built a composite biomarker, which allowed to classify de novo parkinsonian patients against controls (healthy subjects) with an accuracy (defined as the ratio (correctly classified/total) of 82.6%. This study demonstrated for the first time that a common metabolic dysregulation occurs early in either animal models or in PD patients, thus providing an unbiased diagnostic tool as well as major hypothesis for the understanding of the pathophysiology of the disease and the development of innovative therapeutic approaches.

The goal of BIOPARK is to improve the clinical diagnosis of early PD using the blood biomarker.

To this end, the investigators will study whether the biomarker is able to differentiate between patients with PD >5 years and already treated with dopaminergic drugs (thus with a very high diagnostic confirmation) and patients suffering from other neurodegenerative diseases often confused with it, mainly Multiple Systeme Atrophy (MSA). Furthermore, the investigators hope to confirm the preliminary results on a new cohort of de novo patients.

For that aim, they will use the already optimized method for biomarker discovery, i.e. Nuclear Magnetic Resonance (NMR)-based metabolomics on patient serum.

ELIGIBILITY:
Inclusion Criteria:

* Patients with de novo Parkinson's disease, without dopaminergic treatment
* Patients with advanced Parkinson's disease (> 5years) with dopaminergic treatment
* Patients with multiple system atrophy

Exclusion Criteria:

* Patients with deep brain stimulation
* Other neurodegenerative diseases
* patients protected by french law (pregnant or lactating women, prisoners, ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients coming for consultation or admission to day clinic of the neurologic department of the university hospital Grenoble.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
validation of the biomarker in advanced stage PD | 2 years
  The main objective of the project is to evaluate whether classification with the biomarker is consistent with the diagnosis in a cohort of parkinsonian patients with high diagnostic confirmation, i.e. patients treated with L-Dopa for over 5 years

SECONDARY OUTCOMES:
Validation of the biomarker in a new cohort of PD patients | 2 years
  The first secondary objective is to assess whether the biomarker predicts disease in a new cohort of de novo parkinsonian patient
Specificity of the biomarker for PD | 2 years
  The second secondary objective is to assess the specificity of the blood biomarker for the differential diagnosis of PD (early and late stage) by measuring it in a patient population with probable AMS (which is a pathology confounding for PD)
Correlation with MDS-UPDRS | 2 years
  The third secondary objective is to assess, for all patients, whether the classification is consistent with the MDS-UPDRS motor score assessed at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Elena Moro, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

REFERENCES:
- [Background] Mallet D, Dufourd T, Decourt M, Carcenac C, Bossu P, Verlin L, Fernagut PO, Benoit-Marand M, Spalletta G, Barbier EL, Carnicella S, Sgambato V, Fauvelle F, Boulet S. A metabolic biomarker predicts Parkinson's disease at the early stages in patients and animal models. J Clin Invest. 2022 Feb 15;132(4):e146400. doi: 10.1172/JCI146400. PMID 34914634